CLINICAL TRIAL: NCT04586465
Title: Dynamic Positron Emission Tomography/Computed Tomography Evaluated the Response of Neoadjuvant Anti-programmed Cell Death Protein 1 Combination With Chemotherapy for Stage Ⅱa-Ⅲb Non-small Cell Lung Cancer
Brief Title: Dynamic PET/CT Evaluated the Response of Neoadjuvant Anti-PD1 Combination With Chemotherapy for Ⅱa-Ⅲb NSCLC
Acronym: DYNAPET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZDWY.XWK.003
Record Dates: First submitted 2020-10-12; First posted 2020-10-14 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2020-10

CONDITIONS: Non-small Cell Lung Cancer Stage II; Non-small Cell Lung Cancer Stage III; PET/CT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: Dynamic PET-CT compared with RECIST to predict therapeutic response treated with neoadjuvant ICI combined with chemotherapy for stage Ⅱ-Ⅲ NSCLC.
Masking Description: Non
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant ICI combination with chemotherapy for stage Ⅱ-Ⅲ NSCLC (Experimental): Eligible patients with clinical stage Ⅱ-Ⅲ NSCLC will receive dynamic PET-CT before and after 3 cycles neoadjuvant pembrolizumab plus chemotherapy, then patients receive surgical resection. Changes in tumor size were evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. Net uptake rate constant of FDG-Ki value based on dynamic PET will be calculated to evaluate Ki changes before and after treatment. Pathological tumor response were evaluated according to IASLC recommendations. Dynamic PET will be compared with RECIST whether it can better predict the pathological tumor response and disease free survival.
  Interventions: Drug: pembrolizumab, pemetrexed, gemcitabine, cisplatin, carboplatin

INTERVENTIONS:
Drug: pembrolizumab, pemetrexed, gemcitabine, cisplatin, carboplatin — Patients will receive 3 cycles pembrolizumab 200mg, fix dose, 60 minute IV infusion combination with chemotherapy.
  Chemotherapy regimen: ① Eligible patients with non-squamous cell lung cancer, Pemetrexed 500mg/m2, IV infusion on day 1 and cisplatin 75mg/m2 or carboplatin area under the curve (AUC=5), on day 1 of a 3-week schedule for 3 cycles. ② Eligible patients with squamous cell lung cancer. Patients will receive gemcitabine 1250mg/m2 IV on day 1 and day 8, and cisplatin 75mg/m2 or carboplatin AUC=5 on day 1 of a 3-week schedule for 3 cycles
  Other Names: Non

SUMMARY:
The neoadjuvant Immune Checkpoint Inhibitor (ICI) or ICI combination with chemotherapy for Non-small cell lung cancer (NSCLC) had induced higher major pathologic response (MPR) and complete pathological response (PCR). However, the RECIST underestimated the therapeutic response of neoadjuvant ICI therapy. In this study, dynamic PET/CT compared with RECEST 1.1 for the prediction of therapeutic response of NSCLC treated with neoadjuvant ICI combination with chemotherapy.

DETAILED DESCRIPTION:
The prognosis of stage Ⅱa-Ⅲb NSCLC was worse, with 5-year survival rate between 26%-60% after resection. Neoadjuvant ICI or ICI combination with chemotherapy had induced high rate major pathologic response (MPR) and complete pathological response (PCR) for NSCLC. CT image (RECIST) underestimate the response of neoadjuvant therapy. In Checkmate 159 trial, 21 patients with stage Ⅰ-Ⅲa NSCLC received two dose preoperative Nivolumab, only 2 (10%) patients were partial response on CT image assessment. While 9 of 20 (45%) patients were MPR on pathological examination. 2 patients shows tumor progression on CT, but one patient achieved PCR and another patient achieved MPR.Therefore, conventional RECIST criteria cannot accurately assess tumor response to treatment.

The occurrence, development and metastasis of tumor are essentially a series of biochemical processes of abnormal gene expression and metabolism, dysfunction and structural change. 18F-FDG can reflect the metabolic changes of the body at the cellular and molecular level, and the transmission of these metabolic information is earlier than the anatomical changes. By detecting the uptake of 18F-FDG and analyzing tumor metabolism, tissue blood perfusion, receptor, etc., it can provide a theoretical basis for monitoring the therapeutic effect of lung cancer with PET.

As a new imaging technique, 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (18F-FDG) PET/CT is playing an increasingly important role in the diagnosis of tumors. 18F-FDG PET/CT reflects the glucose metabolism process of tumor tissues, and the diagnosis of benign and malignant tumors is based on the difference in glucose metabolism activity between tumor cells and normal tissue cells. 18F-FDG is an isomer of glucose, which is involved in glucose metabolism. Because it is deoxidized and cannot produce hexose bisphosphate, it cannot participate in the next metabolism, and is trapped in cells. In tumor cells, 18F-FDG uptake is increased due to high expression of glucose transport messenger ribonucleic acid (mRNA), elevated glucose transporter Glut-1 and Glut-3 levels, increased hexokinase expression, and down-regulation of glucose-6-phosphatase levels.Molecular imaging using 18F-FDG PET/CT can provide metabolic information to enable better differentiation of benign and malignant tissues and reveal functional abnormalities before structural damage. At the same time, 18F-FDG PET-CT is an effective method for early monitoring of tumor response. It can monitor the metabolic changes of the body before and after tumor treatment, so as to suggest the response of the body to relevant treatment. However, all the PET/CT scans reported in the relevant literature are based on routine static scans, that is, the image data is based on the static images of the tracer obtained at a fixed time point after injection of 18F-FDG. Conventional static PET (60min post-injection scan) can only be used for qualitative visual analysis or semi-quantitative indicator standardized uptake values (SUV) to determine tumor response to treatment. SUV is vulnerable to the influences of uptake time, blood glucose concentration, insulin level, individual weight and injection dose, making it difficult to accurately and quantitatively evaluate tumor response before and after treatment. In order to improve, we plan to adopt dynamic scanning, that is, collecting dynamic data of whole body tissues at all times from the instant of injection of 18F-FDG to one hour. Dynamic scanning can provide information about the temporal metabolism and distribution of the tracer in the tissue, so it can provide more abundant information about the metabolism and distribution of tumor foci and metastasis foci than static scanning, so it can accurately quantify the tumor response before and after treatment. At the same time dynamic PET does not increase the patient's radiation dose compared to static PET.

This study intends to evaluate the efficacy of neoadjuvant anti-programmed cell death protein 1 (anti-PD1) immunotherapy combined with chemotherapy followed by surgery, evaluate the evaluation value of dynamic PET-CT for the efficacy of neoadjuvant therapy, and evaluate the relationship between circulating tumor DNA (ctDNA) changes and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC, performed on a biopsy that occurred within the last 60 days
* Computed tomography (CT) and Dynamic PET-CT within the last 30 days showing radiographic stage Ⅱa to Ⅲb lung cancer (mediastinal staging biopsy is allowed but not required) by the American Joint Committee on Cancer (AJCC) 8th edition
* Potentially surgically resectable by a senior thoracic surgeon
* No driver gene mutation.
* Age≥18 years, and ≤75 years
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the investigator
* Adequate tissue specimens for correlative biomarker analysis. The patient should be willing to provide tissue from a newly obtained biopsy of a tumor lesion and surgical resected tumor lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy or surgical procedures to NCI CTCAE version (v)5.0 grade 1
* Be willing and able to provide written informed consent for the trial
* Absolute neutrophil count (ANC) >= 1500 cells/ microlitre(uL) (within 10 days prior to the start of trial treatment). Platelets >= 100 000 cells/uL (within 10 days prior to the start of trial treatment). Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks) (within 10 days prior to the start of trial treatment). Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance, glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl) >= 30 mL/min for patients with creatinine levels > 1.5 x institutional ULN (within 10 days prior to the start of trial treatment)
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 x ULN (within 10 days prior to the start of trial treatment)
* Aspartate aminotransferase (AST) or serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) or serum glutamate pyruvate transaminase（SGPT) =< 2.5 x ULN (=< 5 x ULN for patients with liver metastases) (within 10 days prior to the start of trial treatment)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 10 days prior to the start of trial treatment)
* Activated partial thromboplastin time (aPTT)/PTT =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 10 days prior to the start of trial treatment)
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of trial medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Male and female patients of childbearing potential must be willing to use an adequate method of contraception as outlined, for the course of the trial through 120 days after the last dose of trial drug o Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient

Exclusion Criteria:

* Any approved anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 5 years prior to initiation of study treatment; however, the following are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Herbal therapy > 1 week prior to Cycle 1, Day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to Cycle 1, Day 1)
* Malignancies other than the disease under study within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score ≤ 6, and prostate-specific antigen (PSA) ≤ 10 mg/mL, etc.)
* Patients who are receiving any other investigational agents concurrently.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab, cisplatin, carboplatin, pemetrexed or gemcitabin.
* Patients with active hepatitis B or C infections or a history of HIV infection.
* Patients with past or resolved hepatitis B infection, defined as having a negative hepatitis B surface antigen (HBsAg) test and a positive for the antibody test to detect antibodies to hepatitis B core antigen (anti-HBc) are eligible.
* Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection including tuberculosis (TB), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1 Received oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study
* Pregnant women
* History of interstitial lung disease or pneumonitis of any cause
* Is ineligible for an operation based on medical or oncologic contraindications to surgery
* Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of trial treatment o Note: Patients who have entered the follow-up phase of an investigational trial may participate as long as it has been 4 weeks after the last dose of the previous investigational agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Major pathological response | up to 12 weeks; analysis of surgical resected tumor samples after neoadjuvant therapy
  10% or less residual viable tumor cells
Dynamic SUV change | up to 12 weeks; analysis change of SUV before and after neoadjuvant therapy
  Dynamic PET-CT SUV change
Objective response rate | up to 12 weeks; analysis change of before and after neoadjuvant therapy
  CT image assessment of tumor response according to RECIST 1.1 criteria
uptake rate constant (Ki) changes | up to 12 weeks; before and after neoadjuvant therapy
  uptake rate constant (Ki) changes before and after neoadjuvant therapy

SECONDARY OUTCOMES:
Progression free survival | up to 3 years
  Time from enrollment to disease progression or death from any cause, whichever occurred first
Treatment related adverse events | 12 weeks
  the number of adverse events related to ICI or platinum-based chemotherapy as evaluated according to CTCAE v4.0.
ctDNA change | 12 weeks
  the amount of ctDNA before and after neoadjuvant therapy

CONTACTS AND LOCATIONS:
Locations (1):
- the fifth affiliated hospital of Sun yat-sen university, Zhuhai, Guangdong, China